CLINICAL TRIAL: NCT02998268
Title: Randomized, Multicenter Phase II Study of Pembrolizumab in Combination With Chemotherapy and Chemoradiation in Locally Advanced Esophageal Adenocarcinoma
Brief Title: Study of Pembrolizumab in Locally Advanced Esophageal Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1602016966
Record Dates: First submitted 2016-11-29; First posted 2016-12-20 (Estimated); Results first posted 2024-05-02 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — pembrolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Other): Subjects in Cohort 1 receive conventional induction chemotherapy with taxol/ carboplatin followed by weekly chemoradiation (taxol/ carboplatin) with pembrolizumab. Following surgery, pembrolizumab is administered every 3 weeks for 1 year.
  Pembrolizumab dosing is 200 mg administered as a 30 minute IV infusion.
  Interventions: Drug: Pembrolizumab; Drug: Taxol; Drug: Carboplatin
- Cohort 2 (Experimental): Subjects in Cohort 2 receive pembrolizumab along with induction chemotherapy with taxol/ carboplatin followed by weekly chemoradiation (taxol/ carboplatin) with pembrolizumab. Following surgery, pembrolizumab is administered every 3 weeks for 1 year.
  Pembrolizumab dosing is 200 mg administered as a 30 minute IV infusion.
  Interventions: Drug: Pembrolizumab; Drug: Taxol; Drug: Carboplatin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Other Names: Keytruda
Drug: Taxol — Taxol is a novel antimicrotubule agent that promotes the assembly of microtubules from tubulin dimers and stabilizes microtubules by preventing depolymerization. This stability results in the inhibition of the normal dynamic reorganization of the microtubule network that is essential for vital interphase and mitotic cellular functions.
  Other Names: Paclitaxel
Drug: Carboplatin — Carboplatin is a platinum coordination compound that is used as a cancer chemotherapeutic agent. Carboplatin produces predominantly interstrand DNA cross-links rather than DNA -protein cross-links.

SUMMARY:
This is a randomized, multicenter phase II study of pembrolizumab in combination with chemotherapy and chemoradiation in locally advanced esophageal adenocarcinoma to examine the safety and efficacy of the combination of pembrolizumab with chemotherapy and chemoradiation in locally advanced esophageal adenocarcinoma as assessed by 1 year disease free survival rate.

DETAILED DESCRIPTION:
This is a randomized, multicenter phase II study of pembrolizumab in combination with chemotherapy and chemoradiation in locally advanced esophageal adenocarcinoma to examine the safety and efficacy of the combination of pembrolizumab with chemotherapy and chemoradiation in locally advanced esophageal adenocarcinoma as assessed by 1 year disease free survival rate. The investigators primary aim is to examine the safety and efficacy of pembrolizumab in both pre-operative treatment paradigms for esophageal/GEJ carcinoma. The specific rationale for the investigators study design is rooted in three unanswered questions:

1. does the addition of an immune check-point inhibitor (pembrolizumab) enhance the efficacy of cytotoxic therapy (chemotherapy with chemoradiation) as determined by response rates, nodal down-staging and 1 year disease free survival in comparison to historical controls,
2. what are the pathological effects of combining pembrolizumab with chemotherapy alone, and
3. what are the molecular (PD-L1 expression), immunological (TILs extent) and gene-expression signatures associated with the efficacy of pembrolizumab in the neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed esophageal or GEJ adenocarcinoma
2. Clinical tumor stage should be T2 Npositive M0 or T3--T4, Nany, M0
3. Be willing and able to provide written informed consent/assent for the trial
4. Be 18 years of age or older on day of signing informed consent.
5. Be a candidate for surgical resection.
6. Be willing to provide tissue during endoscopic assessment of their tumor.
7. Have a performance status of 0 or 1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function as defined below, all screening labs should be performed within 14 days of treatment initiation.

   * Absolute neutrophil count (ANC) ≥1,500 /mcL
   * Platelets≥100,000 / mcL
   * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion within 7 days of assessment
   * Serum creatinine OR Measured or calculated creatinine clearance ≤1.5 X upper limit of normal (ULN) OR
   * ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (Creatinine clearance should be calculated per institutional standard) (GFR can also be used in place of creatinine or CrCl)
   * Serum total bilirubin ≤ 1.5 X ULN OR
   * Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN
   * Albumin >2.5 mg/dL
   * International Normalized Ratio (INR) OR Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
   * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 7 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Evidence of metastatic disease.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has active TB or a history of active TB within 10 years of registration (Bacillus Tuberculosis)
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer treatment, including chemotherapy, radiation, or monoclonal antibody (mAb) for their current diagnosis of esophageal adenocarcinoma.
7. Has a known additional malignancy that is active. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has a previous invasive malignancy treated with curative intent less than 3 years from time of registration. Exceptions include prostate cancer, basal cell squamous skin cancer, and cervical cancer.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2026-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - USC Keck School of Medicine, Norris Cancer Center, Los Angeles, California
  - University of Michigan, Ann Arbor, Michigan
  - Weill Cornell Medicine, New York, New York
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Subjects in Cohort 1 receive conventional induction chemotherapy with taxol/ carboplatin followed by weekly chemoradiation (taxol/ carboplatin) with pembrolizumab. Following surgery, pembrolizumab is administered every 3 weeks for 1 year.
  Pembrolizumab dosing is 200 mg administered as a 30 minute IV infusion.
  Pembrolizumab: Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Taxol: Taxol is a novel antimicrotubule agent that promotes the assembly of microtubules from tubulin dimers and stabilizes microtubules by preventing depolymerization. This stability results in the inhibition of the normal dynamic reorganization of the microtubule network that is essential for vital interphase and mitotic cellular functions.
  Carboplatin: Carboplatin is a platinum coordination compound that is used as a cancer chemotherapeutic agent. Carboplatin produces predominantly interstrand DNA cross-links rather than DNA -protein cross-links.
- Cohort 2: Subjects in Cohort 2 receive pembrolizumab along with induction chemotherapy with taxol/ carboplatin followed by weekly chemoradiation (taxol/ carboplatin) with pembrolizumab. Following surgery, pembrolizumab is administered every 3 weeks for 1 year.
  Pembrolizumab dosing is 200 mg administered as a 30 minute IV infusion.
  Pembrolizumab: Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Taxol: Taxol is a novel antimicrotubule agent that promotes the assembly of microtubules from tubulin dimers and stabilizes microtubules by preventing depolymerization. This stability results in the inhibition of the normal dynamic reorganization of the microtubule network that is essential for vital interphase and mitotic cellular functions.
  Carboplatin: Carboplatin is a platinum coordination compound that is used as a cancer chemotherapeutic agent. Carboplatin produces predominantly interstrand DNA cross-links rather than DNA -protein cross-links.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 20 | 22
Completed | 20 | 19
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Full Range); unit: years] | 61.87 [38.36 to 75.26] | 67.38 [48.22 to 81.96] | 65.06 [38.36 to 81.96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 15 | 18 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 21 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Pathological Response
Description: Tumor tissue will be assessed for major pathological response as defined as complete response or near complete response. Pathologic response was assessed by tumor regression grade. This is a pathologic assessment of the amount of residual cancer cells in the specimen and the degree of fibrosis in the sample specimen. A completer response is 0% residual cancer cells. A partial response is 10-50% residual cancer cells, and no response is >50% residual cancer cells within the tumor specimen.
Time Frame: Between approximately week 15 to 19
Population: 3 participants in Cohort 2 did not have surgery and were therefore ineligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 20 | 19
Participants | 9 | 10

2. Secondary Outcome: R0 Resection Rate.
Description: To examine the efficacy of the combination of pembrolizumab with chemotherapy and chemoradiation as assessed by R0 resection rate, which is reported as the number of participants achieving R0 resection.
Time Frame: 1 year
Population: 1 participant in Cohort 1 and 3 participants in Cohort 2 were unevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 19 | 19
Participants | 17 | 16

3. Secondary Outcome: Overall Survival Rates
Description: To examine the efficacy of the combination of pembrolizumab with chemotherapy and chemoradiation as assessed by overall survival rates
Time Frame: Until death from any cause or for a maximum of 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants That Remained Progression Free as of 1 Year
Description: Number of participants that remained progression free (per RECIST v1.1) and alive as of 1 year
Time Frame: 1 year
Population: 3 participants in Cohort 2 were unevaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 20 | 19
Participants | 15 | 12

5. Other Pre Specified Outcome: Reduction of Local Immune Infiltration.
Description: To explore the effect of the combination of pembrolizumab with chemotherapy as assessed by the local immune infiltration in each treatment group.
Time Frame: Up to 1 year post-surgery
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Prediction of Tumor Response.
Description: To examine whether anti PD1 therapy is associated with a transcriptomic signature of intra-tumoral immune activation predictive of response.
Time Frame: Up to 1 year post-surgery
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Improved 1 Year Survival
Description: To examine whether anti PD1 therapy is associated with a transcriptomic signature of intra-tumoral immune activation predictive of improved 1 year survival.
Time Frame: 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Induction of PD-L1 Expression or Induction of an Inflammatory Signature in Tumors.
Description: To examine whether chemotherapy is associated with induction of PD-L1 expression or induction of an inflammatory signature in tumors
Time Frame: Up to 1 year post-surgery.
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Association of Anti-PD1 Therapy With Increased Intra-tumoral Immune Cell Infiltration.
Description: To examine whether anti PD1 therapy is associated with increased intra-tumoral immune cell infiltration.
Time Frame: Up to 1 year post-surgery.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for a maximum of 30 days from the last dose of study drug administration. The maximum length of time that a participant was followed for AEs is approximately 25 months. Participants are being followed for overall survival for up to 5 years, so mortality data collection is ongoing.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 7/20 | 9/22
Serious Adverse Events (participants affected / at risk) | 8/20 | 13/22
Other Adverse Events (participants affected / at risk) | 20/20 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=20) | Cohort 2 (N=22)
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Bone Infection (Infections and infestations) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cholecystitis (Gastrointestinal disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 — Clostridium difficile
Esophageal anastomotic leak (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0 — Pneumonia
Nausea (Gastrointestinal disorders) | 1 | 2
Neutrophil Count Decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Pleural Infection (Infections and infestations) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Upper Gastrointestinal Bleed (Gastrointestinal disorders) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound Infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=20) | Cohort 2 (N=22)
Abdominal distension (Gastrointestinal disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 16 | 7
Alanine Aminotransferase Increased (Investigations) | 5 | 3
Alkaline Phosphatase Increased (Investigations) | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 13
Anemia (Blood and lymphatic system disorders) | 6 | 9
Anorexia (Metabolism and nutrition disorders) | 12 | 11
Anxiety (Psychiatric disorders) | 3 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 9
Aspartate aminotransferase increased (Investigations) | 5 | 1
Asystole (Cardiac disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Bloating (Gastrointestinal disorders) | 1 | 3
Chills (General disorders) | 2 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 12 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 12
Creatinine Increased (Investigations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 7
Depression (Psychiatric disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 6 | 7
Dizziness (General disorders) | 3 | 3
Dry Skin (Gastrointestinal disorders) | 3 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 12
Dysphagia (Gastrointestinal disorders) | 15 | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Enterocolitis infectious (Infections and infestations) | 2 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 | 5
Esophageal Anastomotic Leak (Injury, poisoning and procedural complications) | 1 | 5
Esophagitis (Gastrointestinal disorders) | 6 | 6
Fatigue (General disorders) | 19 | 18
Fever (General disorders) | 4 | 2
Gait disturbance (General disorders) | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 11 | 0
Generalized muscle weakness (General disorders) | 11 | 6
Headache (Nervous system disorders) | 1 | 2
Hematuria (Renal and urinary disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypertension (Vascular disorders) | 2 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1
Hypotension (Vascular disorders) | 6 | 7
Insomnia (Psychiatric disorders) | 3 | 5
Lung Infection (Infections and infestations) | 1 | 3 — Pneumonia
Lymphocyte count decreased (Investigations) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Nail Infection (Infections and infestations) | 3 | 0
Nausea (Gastrointestinal disorders) | 17 | 11
Neutrophil Count Decreased (Investigations) | 8 | 4
Non-cardiac chest pain (Cardiac disorders) | 5 | 3
Other, atrial arrhythmia (Cardiac disorders) | 5 | 3
Other: Cold Intolerance (General disorders) | 3 | 1
Other: Fungal Infection (Infections and infestations) | 2 | 0
Other: Laryngeal nerve injury (Injury, poisoning and procedural complications) | 0 | 4
Other: Mucositis (Gastrointestinal disorders) | 3 | 0
Other: Rash (Skin and subcutaneous tissue disorders) | 3 | 20
Palpitations (Cardiac disorders) | 0 | 2
Paresthesia (Nervous system disorders) | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 11
Platelet Count Decreased (Investigations) | 3 | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0
Sinus Tachycardia (Cardiac disorders) | 5 | 4
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Syncope (Nervous system disorders) | 0 | 7
Thromboembolic event (Vascular disorders) | 1 | 2
Urinary Tract Infection (Infections and infestations) | 3 | 7
Vomiting (Gastrointestinal disorders) | 11 | 9
Weight Loss (Investigations) | 11 | 12
White blood cell decreased (Investigations) | 3 | 2
Wound infection (Infections and infestations) | 5 | 6
Confusion (Psychiatric disorders) | 3 | 0
Other: Night Sweats (General disorders) | 2 | 0
Pain (General disorders) | 7 | 3
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 2
Edema Limbs (General disorders) | 3 | 2
Other: Increased urinary frequency (Renal and urinary disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 4
Blurred Vision (Eye disorders) | 2 | 0
Other: Myelosuppression (Blood and lymphatic system disorders) | 0 | 3
Other: Odynophagia (Gastrointestinal disorders) | 0 | 2
Other: Shingles (Infections and infestations) | 0 | 2
Other: Hiccups (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT02998268/Prot_SAP_000.pdf